CLINICAL TRIAL: NCT01793220
Title: Economic and Clinical Outcomes of Attendance in Psychosis Services Using SMS: The ECO APSS Randomized Controlled Trial
Brief Title: Economic and Clinical Outcomes of Attendance in Psychosis Services Using SMS.
Acronym: ECO APSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Daniel Hayes, Mr, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ECOAPSS1
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Reminder (Experimental): A text message reminder service will be sent 7 and 1 days(s) prior to the patients appointment at their Psychosis Community Service.
  Interventions: Other: SMS reminder
- No SMS Reminders (No Intervention): The service user will not be sent text message reminders prior to each appointment at their Psychosis Community Service

INTERVENTIONS:
Other: SMS reminder — A text message reminder service will be sent 7 and 1 days(s) prior to the patients appointment at their Psychosis Community Service.
  Arms: SMS Reminder

SUMMARY:
The aim of this research is to find out if mobile phone text message reminders of appointments can help to address missed appointments in Psychosis Community Services. Another aim is to examine if fewer missed appointments result in clinical benefits for service users and in lower costs for Psychosis Community Services over a period of 6 months. 600 users from 2 London Psychosis Community Services will take part in this research. Each participant will be put into one of two groups, as s/he joins the study: In the first (experimental) group, each participant will receive appointment reminders for 6 months (7 and 1 day/s before each appointment), starting with the first available opportunity upon joining the study. In the second (control) group, each participant will not receive appointment reminders for 6 months. The choice of group for each individual will be made at random by a computer. Clinical information will be collected for 6 months from the time each participant joins the study, using, with his or her consent, their anonymised electronic medical records. The following clinical information will be compared between the experimental and control groups: Attendance of appointments, number of inpatient admissions, number of days in inpatient care, number of inpatient admissions under the mental health treatment act, number of referrals to a home treatment team, number of times patient has changed medication, health and social functioning. Service use, service costs and the cost-effectiveness of the reminder system will also be examined. Towards the end of their participation, service users, as well as mental health professionals, will be invited to express their views, concerns and suggestions in relation to the reminder service by completing a brief anonymised (service users) or anonymous (staff) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Be a user of Psychosis Community Services
* Manifest at least a basic level of comprehension of the study (including its nature, purpose, procedures and implications) prior to enrollment, and adequate capacity to consent, as assessed by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) scale.
* Own a mobile phone.
* Be willing to receive SMS reminders of appointments with the Psychosis Community Service.
* Provide written informed consent to participate in the study.

Exclusion Criteria:

* Is not a user of Psychosis Community Services.
* Cannot manifest at least a basic level of comprehension of the study (including its nature, purpose, procedures and implications) prior to enrollment, and/or adequate capacity to consent, as assessed by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) scale.
* Does not own a mobile phone.
* Is under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Outcome of appointment (attended, missed, cancelled by the participant, cancelled by the service) | From baseline to end of intervention (6 months)
  To assess differences in appointment attendance using online patient records in those who receive the SMS appointment reminders and those that do not

SECONDARY OUTCOMES:
Economic outcome: Use of Psychosis Services and impact on cost | From baseline to end of intervention (6 months)
  Data on the use of services over the follow-up period will be combined with appropriate unit cost information (Curtis, 2011; Department of health, 2012). Service costs will be compared between the experimental (SMS intervention) and control (No SMS intervention)groups. Cost data often follow a skewed distribution and so bootstrap methods will be employed
Clinical outcome: Number of inpatient admissions | From baseline to end of intervention (6 months)
  To assess differences in the number of inpatient admissions using online patient records in those who receive the SMS appointment reminders and those that do not
Clinical outcome: Number of days in inpatient care | From baseline to end of intervention (6 months)
  To assess differences in number of days in inpatient care using online patient records in those who receive the SMS appointment reminders and those that do not
Clinical outcome: Number of inpatient admissions under the mental health treatment act | From baseline to end of intervention (6 months)
  To assess differences in number of inpatient admissions under the mental health act using online patient records in those who receive the SMS appointment reminders and those that do not
Clinical outcome: Number of referrals to a home treatment team | From baseline to end of intervention (6 months)
  To assess differences in the number of times a patient has been referred to a home treatment team, using online patient records (a crisis team who further support those with declining mental health) in those who receive the SMS appointment reminders and those that do not
Clinical outcome: Number of times patient has had changes to their medication | From baseline to end of intervention (6 months)
  To assess differences in the number of times patient has had changes to their medication using online patient records in those who receive the SMS appointment reminders and those that do not
Clinical outcome: Level of health and social functioning, as reflected in the patient's score on the Health of the Nation Outcome Scales (HoNOS) | Baseline and 6 months
  To assess differences in levels of health and social functioning in those who receive the SMS appointment reminders and those that do not
Economic outcome: cost effectiveness of the SMS intervention | 1 year after baseline
  The cost of the actual intervention will be negligible given the extent of general SMS use. However, there could be an impact on service costs and this will be estimated. Data on the use of services over the follow-up period (see below for details) will be combined with appropriate unit cost information (Curtis, 2011; Department of health, 2012). Cost-effectiveness will be assessed by combining the cost data with HoNOS scores using an incremental cost-effectiveness ratio. Uncertainty around the cost-effectiveness estimates will be explored using cost-effectiveness planes and cost-effectiveness acceptability curves.

OTHER OUTCOMES:
Views and suggestions of services users in relation to the SMS reminders | 6 months (end of study participation)
  At the end of their participation, service users will be invited to complete an optional brief questionnaire (designed for the purposes of the study by the research team), to express their views, concerns and suggestions in relation to the SMS service. This information will be collected in an anonymised format. The questionnaires will be posted to the study participants, or alternatively, administered to them over the telephone or in person (whichever they prefer) by a research worker.
Views and suggestions of mental health professionals in relation to the SMS reminders | After the study has ended (1 year after 1st recruitment)
  At the end of ths study, staff from participating services will be invited to complete an optional brief questionnaire (designed for the purposes of the study by the research team), to express their views, concerns and suggestions in relation to the SMS service. This information will be collected in an anonymous format. The questionnaires will be given to staff and posted back to the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Hayes, MSc, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, Greater London, United Kingdom